CLINICAL TRIAL: NCT03582748
Title: Neuroimaging Predictors of Bariatric Surgical Outcome
Status: Active, not recruiting | Type: Observational
Sponsor: Hartford Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: HHC-2017-0147
Record Dates: First submitted 2018-06-14; First posted 2018-07-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- New surgical subjects: This group will be consist of 150 consecutively consented subjects who are scheduled to have sleeve gastrectomy at the Hartford Hospital Surgical Weight Loss Center.
  Interventions: Procedure: sleeve gastrectomy
- Carry over surgical subjects: This group will include 45 subjects who participated in the pilot study and who will be contacted and consented into the present study.
  Interventions: Procedure: sleeve gastrectomy
- Non-surgical subjects: This group will include 15 non-surgical patients who will be group-matched to Group A on pertinent characteristics. These patients will be non-surgical in that they will have been evaluated for bariatric surgery by the SWLC but deemed ineligible for any of a number of reasons.
  Interventions: Procedure: No sleeve gastrectomy

INTERVENTIONS:
Procedure: sleeve gastrectomy — removal of most of stomach as a bariatric surgical procedure
  Groups: Carry over surgical subjects; New surgical subjects
Procedure: No sleeve gastrectomy — Non-receipt of sleeve gastrectomy procedure
  Groups: Non-surgical subjects

SUMMARY:
Bariatric surgery is an important treatment option for morbidly obese patients who fail to lose weight through diet and exercise. Despite intervention, 20-50% of patients either fail to lose targeted amounts of weight or regain weight that was lost initially. Attempts at predicting degree of weight loss have had only modest success and none have long term (>2 year) reliability. Moreover, research predicting weight loss beyond the 1st or 2nd year post-surgery and for outcomes other than weight loss including comorbidities common in the bariatric population is lacking. The investigators' pilot data in 45 patients suggest that individual differences on pre-surgical neural activity measured with functional MRI (fMRI) reliably explains 33% of the variance in weight loss up to 1 year post surgery, and over 50% of a multifaceted outcome measure, far outperforming many other indicators. These predictors implicate regions that closely conform to a theoretical model emphasizing both consummatory urges (a "Now" neural circuit) vs. regulation of craving and self-control (a "Later" circuit). The central hypothesis in this study is that individual differences in these neural pathways exert a powerful effect on the ability to sustain weight loss and achieve other key health outcomes.

The study will replicate and refine this model over a longer timeframe and assess its predictive utility for key weight-related health outcomes. The investigators propose to replicate the model derived from their fMRI pilot data and secondarily to explore its predictive utility for changes in calorie intake, activity levels, liver fat, hemoglobin A1c, plasma lipids, blood pressure, and fasting glucose in a new, independent cohort of N=150 successively consenting, presurgical sleeve gastrectomy (SG) patients in study years 1-3. The study will follow the pilot cohort for up to 7 years and the new cohort for 3 or more years to determine if predictors replicated in Aim 1 retain their long-term predictive power, particularly when supplemented with non-brain imaging variables and using a larger longitudinal dataset. The study will use imaging and non-imaging data to develop multivariate statistical models incorporating energy balance, fMRI, and laboratory values with the variables described in Aim 1 to help to separate predictors vs. consequences of post-surgical outcomes. To help separate scan-to-scan variability from true post-surgical, trajectory-related brain changes, the study will enroll N=20 obese subjects who will not undergo bariatric surgery, and are individually matched with the above SG subjects. Finally, the study will evaluate whether several related, non-fMRI cognitive tests might potentially act as surrogates in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Right handed
* Scheduled to undergo sleeve gastrectomy at the Hartford Hospital Surgical Weight Loss center (new surgical subjects)
* able to understand purpose of study as presented in English

Exclusion Criteria:

1. Auditory or visual impairment that interferes with test-taking.
2. Mental retardation (WAIS Full Scale IQ<70).
3. Traumatic brain injury with loss of consciousness > 10 minutes or concussion in last 20 days.
4. Presence or history of any medical/neurologic illness that may affect brain physiology (e.g., epilepsy, multiple sclerosis), including focal brain lesion seen on structural MRI (all structural scans are read by a licensed radiologist).
5. Current pregnancy (all pre-menopausal females (i.e., those still having menstrual periods) will be tested with urine screens on the day of MRI).
6. Presence of marijuana, cocaine, opiates, alcohol or substance dependence. All participants will receive a urine screen for the presence of marijuana, cocaine, opiates and a breath screen to detect the presence of alcohol. Any positive substance screen will result in exclusion. Subjects with substance dependence will be excluded, including those dependent on caffeine and nicotine based on psychiatric interviews and instruments such as the Fagerstrom Test of Nicotine Dependence
7. Any tobacco use.
8. Current or lifetime SCID Axis I DSM-IV-TR psychotic disorder diagnosis, substance abuse/dependence diagnosis or report of psychotic disorder in a first-degree relative.
9. Inability to understand spoken English sufficiently to comprehend testing procedures available in English, inability to speak English fluently (or is non-native English speaker or was educated in a primary language other than English past grade 1).
10. Inability to comprehend the consent form appropriately.
11. Other specific fMRI exclusions, including metal devices, clips or fragments in body.
12. Body weight > 550 lb (due to the weight restrictions of the MRI table).
13. Left handedness.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Bariatric surgery patients who have elected to receive sleeve gastrectomy (SG) surgery or who were pursuing SG but were not candidates for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Body weight | up to 7 years

SECONDARY OUTCOMES:
Regulation of Craving (ROC) functional MRI (fMRI) Task | up to 7 years
  This task tests food cue- induced craving and the ability to regulate craving. Participants are given an instruction, see pictures of high-calorie foods (previously shown to increase craving) and then rate their craving on a scale from 1 (not at all) to 5 (a lot).
Monetary Incentive Delay Task (MID) fMRI Task | up to 7 years
  Participants see cues that they may win or lose money ($0, $1, $5), then wait for a variable anticipatory delay period, and respond to a rapidly presented target with a single button press to try to either win or avoid losing money.
Affective Pictures Paradigm (APP) fMRI Task | up to 7 years
  This task examines neural activity elicited by incidental emotional processing that engages emotional systems. Forty-two single-face pictures (14 happy, 14 angry and 14 neutral expressions) are presented in pseudorandom order for 3 sec with a 9-sec inter-stimulus interval during which a fixation cross serves as a baseline measure. Participants are instructed to identify via button press whether the face was male or female.

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No